CLINICAL TRIAL: NCT07248722
Title: Effect of Acid-suppression Drugs on Short-term Outcomes After Prophylactic Endoscopic Variceal Treatment in Cirrhosis: A Multicenter Randomized Controlled Trial
Brief Title: Acid-suppression Drugs After Prophylactic Endoscopic Variceal Treatment of Esophagogastric Variceal Bleeding in Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XHNKKY-EVT-ASD
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Esophageal and Gastric Varices; Liver Cirrhosis
Keywords: esophageal and gastric varices; endoscopic therapy; acid suppression; adverse events; liver cirrhosis
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD group (Experimental)
  Interventions: Drug: ASD
- non-ASD group (No Intervention)

INTERVENTIONS:
Drug: ASD — Patients should receive intravenous esomeprazole 40 mg/d immediately after EVT for 3 to 7 days until discharge, followed by oral keverprazan 20 mg/d until the total duration of acid suppression is 2 weeks.
  Other Names: acid-suppression drugs
  Arms: ASD group

SUMMARY:
Traditionally, it is considered that gastric acid delays ulcer healing, and acid suppression can reduce the risk of post-banding ulcer bleeding and promote mucosal healing at the ulcer site. A systematic review and meta-analysis performed by our team demonstrated that acid suppression significantly reduced the incidence of bleeding following prophylactic endoscopic variceal treatment (EVT), but had no significant effect on the incidence of mortality, adverse events, or length of stay. Similarly, another systematic review and meta-analysis performed by Lin et al. indicated that PPIs significantly reduced the incidence of bleeding after therapeutic or prophylactic EVT, and the efficacy of PPIs in reducing post-EVT bleeding is related to the duration of PPIs. However, previous studies have indicated that long-term use of acid-suppression drugs (ASD) may increase the risk of bacterial infections and hepatic encephalopathy in patients with cirrhosis. Therefore, current guidelines suggest that ASD should be discontinued after EVT, unless the patient has a clear indication for acid suppression. However, the quality of evidence is poor due to the small sample sizes, predominantly retrospective designs, and inconsistencies in follow-up duration of previous studies. In current clinical practice, most physicians still prefer to use ASD routinely after EVT to prevent post-EVT bleeding. Given the ongoing controversy regarding the routine use of ASD after EVT, we plan to conduct a multicenter randomized controlled trial to evaluate the effects of the use of ASD after prophylactic EVT on short-term bleeding, adverse events, and mortality in patients with cirrhosis.

DETAILED DESCRIPTION:
Overall, 210 patients with cirrhosis undergoing prophylactic EVT will be enrolled. They will be randomly assigned at a ratio of 1:1 to the ASD group and non-ASD group. The primary endpoint is 6-week bleeding. Secondary endpoints include 6-week all-cause mortality and adverse events (retrosternal pain/discomfort, nausea/vomiting, heartburn/acid regurgitation, fever, diarrhea, abdominal pain, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of liver cirrhosis confirmed by liver biopsy and/or a combination of clinical manifestation, laboratory, and imaging examinations;
2. endoscopically confirmed esophagogastric varices and undergoing EVT;
3. patients aged ≥18 years, regardless of gender;
4. sign the informed consent form.

Exclusion Criteria:

1. diagnosis of acute upper gastrointestinal bleeding upon admission, with clinical manifestations such as hematemesis, melena, and/or hematochezia;
2. definite indications for acid suppression upon admission: reflux esophagitis, peptic ulcer, Zollinger-Ellison syndrome, etc.;
3. definite indications for acid suppression discovered during EVT: reflux esophagitis, peptic ulcer, etc.;
4. allergy to ASD or previous intolerable adverse reactions to ASD;
5. severe cardiovascular or cerebrovascular diseases or renal impairment;
6. severe hematological disorders;
7. women preparing for pregnancy or those who were pregnant and lactating;
8. patients who have already participated in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of 6-week bleeding | 6 weeks

SECONDARY OUTCOMES:
Rate of 6-week all-cause mortality | 6 weeks
Rate of 6-week adverse events | 6 weeks
  retrosternal pain/discomfort, nausea/vomiting, heartburn/acid regurgitation, fever, diarrhea, abdominal pain, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, Study Director — Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area)
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin L, Cui B, Deng Y, Jiang X, Liu W, Sun C. The Efficacy of Proton Pump Inhibitor in Cirrhotics with Variceal Bleeding: A Systemic Review and Meta-Analysis. Digestion. 2021;102(2):117-127. doi: 10.1159/000505059. Epub 2020 Feb 21. PMID 32088712
- [Result] Zhang YY, Wang L, Shao XD, Zhang YG, Ma SZ, Peng MY, Xu SX, Yin Y, Guo XZ, Qi XS. Effects of postoperative use of proton pump inhibitors on gastrointestinal bleeding after endoscopic variceal treatment during hospitalization. World J Gastrointest Surg. 2023 Jan 27;15(1):82-93. doi: 10.4240/wjgs.v15.i1.82. PMID 36741070
- [Result] Zhu J, Qi X, Yu H, Su C, Guo X. Acid suppression in patients treated with endoscopic therapy for the management of gastroesophageal varices: a systematic review and meta-analysis. Expert Rev Gastroenterol Hepatol. 2018 Jun;12(6):617-624. doi: 10.1080/17474124.2018.1456918. Epub 2018 Apr 4. PMID 29564926